CLINICAL TRIAL: NCT01597102
Title: Cerebrovascular Autoregulation During and After Liver Transplantation
Acronym: dARICULtx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, Principal investigator, Johannes Gutenberg University Mainz
Other Study IDs: 837.041.10 III
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Encephalopathy, Hepatic; Cerebrovascular Disorders; Liver Failure
Keywords: encephalopathy, hepatic; autoregulation, cerebrovascular; liver failure; liver transplantation
MeSH Terms: conditions — Hepatic Encephalopathy; Cerebrovascular Disorders; Liver Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver transplantation: Patients with liver failure and liver transplantation
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No intervention is planned in this study
  Other Names: No intervention is planned in this study

SUMMARY:
The cerebrovascular autoregulation (AR) is impaired in patients with hepatic encephalopathy. Patients with the indication to liver transplantation mostly have mild to severe hepatic encephalopathy. Transplantation should recover the encephalopathy. The aim of the study is to investigate the AR during liver transplantation, with the questions if the AR is impaired at the beginning of surgery and if there are changes in AR. For follow up the AR will be measured at the first days after transplantation at the ICU.

DETAILED DESCRIPTION:
The cerebrovascular autoregulation (AR) will be measured using transcranial doppler and calculating the index of autoregulation Mx. This measurement is continuous with online calculation. So, the possible changes over the whole time of surgery can be detected. Furthermore, the measurement of AR at the ICU will be performed daily at the same time over a measurement period of 60 Minutes and the time course of AR after liver transplantation will be described.

ELIGIBILITY:
Inclusion Criteria:

* liver transplantation
* age > 18 years

Exclusion Criteria:

* sepsis
* preexisting cerebral diseases
* traumatic brain injury
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with and stage liver failure and transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-01-08 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes of cerebrovascular autoregulation during liver transplantation | During the surgery
  Measuring cerebrovascular autoregulation during the whole liver transplantation and compare the index of AR at the beginning with index of AR Mx after reperfusion of the transplantated liver

SECONDARY OUTCOMES:
Time course of cerebrovascular autoregulation after liver transplantation | First 4 days after transplantation
  Meaurement of cerebrovascular autoregulation daily for the first 4 days and calculating a time course

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schramm, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- University Medical Center, Mainz, Germany